CLINICAL TRIAL: NCT06526416
Title: Anterior Chamber Angle Changes After Bent Angle Needle Goniectomy Procedure, Anterior Segment OCT Study
Brief Title: The Objective is to Evaluate the Anterior Chamber Angle After BANG Procedure, the Study Will Recruit 12 Patients Who Will Undergo Planned Goniectomy for Uncontrolled POAG, Anterior Segment OCT Scan Will Be Used to Evaluate the Anterior Chamber Postoperatively.
Status: Not yet recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Nader Hussein Fouad Hassan, Lecturer in Ophthalmology, Benha University
Other Study IDs: RC.50.5.2023
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Primary Open Angle Glaucoma; Glaucoma
Keywords: Bent angle needle goniectomy; anterior segment optical coherence tomography; Primary open angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Anterior segment optical coherence tomography — Imaging of the anterior segment of the eye using optical coherence tomography

SUMMARY:
Evaluation of anterior segment using anterior segment optical coherence tomography in patients undergoing planned bent angle needle goniectomy procedure for uncontrolled open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are being treated for primary open angle glaucoma using eye drops.
2. Patients with uncontrolled intraocular pressure >21 mm Hg
3. All recruited patients should have open anterior chamber angles demonstrated on gonioscopy examination.
4. Patients giving consent for operation and follow up

Exclusion Criteria:

* 1- Pseudophakic patients 2- Advanced glaucoma patients. 3- Patients who are to have trabeculectomy or laser trabeculoplasty. 4- Patients with secondary glaucoma. 5- Patients who are unable to give consent for surgery or follow up. 6- Patients with previous trauma to the eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients presenting to Benha University Hospitals with open angle glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To detect the changes in anterior chamber angle using Anterior segment OCT after BANG goniectomy | 12 weeks after the day of surgery.
  To detect the changes in anterior chamber angle using Anterior segment OCT after BANG goniectomy

SECONDARY OUTCOMES:
To detect any correlation between the post-op anterior chamber angle changes and the intraocular pressure. | 12 weeks after the day of surgery.
  To detect any correlation between the post-op anterior chamber angle changes and the intraocular pressure.